CLINICAL TRIAL: NCT05867173
Title: Development and Assessment of Listener-tailored Programming for Cochlear Implant Listeners
Brief Title: Perceptual Consequences of Cochlear Implant Electrode-neuron Interfaces
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Boston Children's Hospital (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Julie G. Arenberg, CCC-A, Director of Research and Education, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: MGB_2019P000239
Record Dates: First submitted 2023-02-27; First posted 2023-05-19 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Performance Assessed with Experimental Sound Processing Strategy (Experimental): Patients listening to experimental cochlear implant processing strategy.
  Interventions: Other: Experimental Speech Processing Strategy
- Control (No Intervention): Patients listening to their clinical cochlear implant using their "own" processor (their everyday listening situation).
- Experimental Control (Sham Comparator): Patients listening to experimental cochlear implant using a processing strategy like thier clinical program, a "clinical like" program.
  Interventions: Other: Experimental Speech Processing Strategy

INTERVENTIONS:
Other: Experimental Speech Processing Strategy — Patient's will listen with an experimental speech processor, programmed with a dynamic focusing strategy.
  Arms: Experimental Control; Performance Assessed with Experimental Sound Processing Strategy

SUMMARY:
Despite the success of cochlear implants, devices surgically placed in the inner ears of patients with severe hearing loss, there remains substantial variability in the overall speech perception outcomes for the children and adults who receive them. The main goals of this project are: i) to improve our understanding of how cochlear implants affect the developing auditory system, ii) apply that knowledge to test new methods for programming children and adults, and iii) to study how long it takes listeners to adapt to new cochlear implant programs over the short- and long-term. The results will improve our understanding of how the deafened auditory system develops with cochlear implant stimulation and advance clinical practice to improve hearing outcomes in cochlear implant listeners.

ELIGIBILITY:
Inclusion Criteria:

Research Subjects with a Cochlear Implant ADULTS Inclusion Criteria

* Adult at least 18 years old
* Native speakers of American English
* Wears a cochlear implant manufactured by Advanced Bionics (Clarion Hi-Focus I or newer), Cochlear, or MED-EL

CHILDREN Inclusion Criteria

* Children at least 3 months old
* Native speakers of American English
* Wears a cochlear implant manufactured by Advanced Bionics (Clarion Hi-Focus I or newer), Cochlear, or MED-EL

  * For both children and adults with a cochlear implant, some study criteria might pertain to a subset of subjects, such as a specific age at which the subjects developed a hearing loss, or was implanted.

Exclusion Criteria:

Exclusion for all Cochlear Implant Subjects:

* Inability to provide informed consent
* Does not meet the inclusion criteria for a specific study protocol, such as age of onset of hearing loss, age of cochlear implantation, duration of deafness, number of active electrodes in the cochlear implant device
* Unable to carry out the study protocol or tasks required in the study

Exclusion for all Normal Hearing Subjects:

* Inability to provide informed consent
* Hearing loss, or significant history of hearing related issues
* Unable to carry out the study protocol or tasks required in the study

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Slopes of the spread of excitation of the electrically evoked compound action potential responses | Baseline
  Responses of the auditory nerve can be measured directly from the cochlear implant using software developed by the implant manufacturer. By changing the distance between two electrodes, we can quantify the spread of activation in the cochlea.
Slopes of a behavioral measure of spectral resolution called psychophysical tuning curves. | Baseline
  A behavioral test designed to measure how spectral information is processed in the auditory system. By changing the relationship between a masker and target signal, we can assess resolution.
Changes in vowel identification scores | Baseline and weekly for 10 weeks after the intervention
  Medial vowel identification performance in background noise. Participants will complete age-appropriate testing.
Changes in sentence recognition scores | Baseline and weekly for 10 weeks after the intervention
  Speech perception testing includes sentence recognition in noise. Participants will complete age-appropriate testing.
Changes in speech-gap detection thresholds | Baseline and weekly for 10 weeks after the intervention
  Speech perception testing includes speech-gap detection. Participants will complete age-appropriate testing.
Changes in phoneme discrimination scores | Baseline and weekly for 10 weeks after the intervention
  Speech perception testing includes phoneme discrimination. Participants will complete age-appropriate testing.
Changes in time (weeks) with programming strategy | Baseline and weekly for 10 weeks after the intervention
  Outcome measures will be obtained at weekly intervals during the intervention, and the weekly collection of those measures will be analyzed.

SECONDARY OUTCOMES:
Age | Age at baseline
  A secondary age analysis on all outcome measures will be applied.
Infant-Toddler Meaningful Auditory Integration Scale (ITMAIS) scores | Baseline, and weekly for 10 weeks after the intervention
  The IT-MAIS is a study-team-guided parental report about how infants and toddlers are responding to sound.
Macarthur-Bates vocabulary inventory scores | Baseline, and weekly for 10 weeks after the intervention
  This test allows the study team and parents to monitor speech and language development, specifically new word learning.
Hearing quality of life (HEARQL) scores | Baseline, 5 weeks, and 10 weeks after the intervention
  The HEAR-QL is a self-assessment test normed for children to assess how they hear in everyday life with different interventions
Sound quality questionnaire | Baseline and weekly for 10 weeks after the intervention
  Participants will be asked to rate sound quality with different interventions in comparison to their everyday listening on a 7-point scale (from minus 3 - much worse, up to plus 3 - much better, 0 is the same)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Arenberg, Principal Investigator — Massachusetts Eye and Ear
Locations (2):
- United States (2):
  - Mass Eye and Ear, Boston, Massachusetts
  - Boston Children's Hospital, Waltham, Massachusetts